CLINICAL TRIAL: NCT06618521
Title: Effect of Pilates Exercise Versus Circuit Exercise Training on Gestational Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Hamed Ibrahim ElMorsy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004254
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gestational Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Antihypertensive Agents; Methyldopa; Exercise Movement Techniques; Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anti-hypertensive drug (Active Comparator): It consists of 23 pregnant women. They will take Anti-hypertensive drug (Methyldopa 250 mg according to physician instructions).
  Interventions: Drug: Anti-hypertensive drug (Methyldopa 250 mg)
- Anti-hypertensive drug + Pilates exercise (Experimental): It consists of 23 pregnant women. They will be engaged in Pilates exercise for 40 minutes/day, 3 days/week, for 12 weeks, in addition to Anti-hypertensive drug (Methyldopa 250 mg according to physician instructions.
  Interventions: Drug: Anti-hypertensive drug (Methyldopa 250 mg); Other: Pilates exercise
- Anti-hypertensive drug + Circuit exercise training (Experimental): It consists of 23 pregnant women. They will be engaged in a supervised circuit training exercises for 40 minutes/ day, 3 days/week, for 12 weeks, in addition to Anti-hypertensive drug (Methyldopa 250 mg according to physician instructions.
  Interventions: Drug: Anti-hypertensive drug (Methyldopa 250 mg); Other: Circuit exercise training

INTERVENTIONS:
Drug: Anti-hypertensive drug (Methyldopa 250 mg) — Each women in the three groups will receive Medical treatment Anti-hypertensive drug (Methyldopa 250 mg) according to physician instructions.
  Other Names: Methyldopa 250 mg
Other: Pilates exercise — Each women in the second group will receive Mat Pilates training exercise for 40 minutes/ day, 3 days/week, for 12 weeks beginning 20 weeks' gestation. The Pilates exercise includes pelvic floor exercise, deep tummy strengthening, pelvic tilt, upper back stretch, the cat stretch, thigh stretch, the sword, sword arm, and wagging the tail.
  Arms: Anti-hypertensive drug + Pilates exercise
Other: Circuit exercise training — Each women in group C will receive circuit training exercises in form of single leg curl up and press, sumo squat and row to reverse fly stand for 40 minutes/ day, 3 days/ week, for 12 weeks beginning 20 weeks' gestation. The Circuit exercise training includes sumo squat, quadruped extension, row to reverse fly stand, and single leg curls up.
  Arms: Anti-hypertensive drug + Circuit exercise training

SUMMARY:
The purpose of the study is to investigate the effect of Pilates exercises versus circuit exercise training on blood pressure and lipids in gestational hypertensive women.

DETAILED DESCRIPTION:
Gestational hypertension is one of the most common disorders seen in human pregnancies. The disorder progresses into pre-eclampsia, a dangerous condition that can prove fatal to expectant mothers. If it is untreated several complications result such as eclampsia, stroke, the need for labor induction and placental abruption, preterm delivery, and low birth weight.

Most pregnant women use medication during pregnancy despite increasing availability of information about teratogenic risks. Medication use during pregnancy still causes uncertainty and concern among pregnant women and their health care providers. Medication use has a harmful effect on the fetus such as congenital anomalies, preterm birth, low birth weight, growth retardation of the fetus, and developmental delays in totality. It remains unknown what the major concerns are among pregnant women regarding medication use.

Health organizations recommend lifestyle changes that include increased levels of physical activity. Also, some researchers have recommended aerobic training for 30 minutes per day that is supplemented with resistance exercise.

Pilates exercises have been showed to be safe modality for pregnant women. It showed many benefits on childbirth. It also yields a significant decrease in clinical systolic and diastolic and mean blood pressure at rest and over 24 hours, in hypertensive non-pregnant women. Pilates may be recommended as a non-drug intervention for the prevention, treatment, and control hypertension. Circuit exercise training is also a non-drug intervention may reduce systemic arterial hypertension to lower cardiovascular risk.

Due to the progressive increase in maternal estrogen with pregnancy, maternal fat deposits switch from anabolic to catabolic states to maintain appropriate development of the fetus and placenta. This switch to catabolism increases the breakdown of fat stores, which increases total cholesterol and triglyceride available for maternal and fetal utilization. Further, it is essential for a normalized maternal lipid profile to ensure healthy fetal development and pregnancy outcomes.

Therefore, this study will be conducted to provide evidence based for the effectiveness of Pilates exercise and circuit training on blood pressure and lipid profile in gestational hypertensive women for healthcare providers interested in women's health.

ELIGIBILITY:
Inclusion Criteria:

* They will be diagnosed by obstetrician after 20 weeks' gestation as having blood pressure higher than 140/90 without any organ damage.
* Age will range from 25-35 years old .
* Body mass index (BMI) will range from 30-34.9 Kg/m².

Exclusion Criteria:

* Cardiac problems
* Cognitive problems
* Poorly controlled hypertension
* Diabetes mellitus
* Inflammatory stage of arthritis
* Osteoporosis

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 69 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Measurement of mean arterial blood pressure | 12 weeks
  Pregnant women will be seated in a relaxed position with the arm supported on a table. A cuff will be secured around the bicep without excessive tightness. The cuff will be inflated while observing the aneroid monitor until the pressure reaches 20-30 mmHg above the usual blood pressure. A stethoscope will be placed below the cuff at the elbow crease, and the cuff will be gradually deflated. Systolic pressure will be recorded at the first Korotkoff sound, and diastolic pressure will be recorded when the sounds disappear. Mean arterial blood pressure will be measured for each pregnant woman in the three groups before and after the treatment procedures using the equation: MAP = 1/3 (SBP) + 2/3 (DBP).
Assessment of serum triglycerides level | 12 weeks
  It will be assessed for each pregnant women in the three groups before and after the end of the treatment procedures.The blood samples will be collected after fasting for 9-12 hours. Participants will be asked to lie in half lying position with well supported back and arm, the antecubital area will be cleaned with alcohol. Blood sample of about 5cm will be drawn in the morning (at 8 clock) range between 7and 25 micrograms per deciliter (mcg-dl). Blood sample will be using disposable syringe and collected in sterilized tube.
Assessment of serum total cholesterol level | 12 weeks
  It will be assessed for each pregnant women in the three groups before and after the end of the treatment procedures.The blood samples will be collected after fasting for 9-12 hours. Participants will be asked to lie in half lying position with well supported back and arm, the antecubital area will be cleaned with alcohol. Blood sample of about 5cm will be drawn in the morning (at 8 clock) range between 7and 25 micrograms per deciliter (mcg-dl). Blood sample will be using disposable syringe and collected in sterilized tube.
Assessment of serum low-density lipoprotein (LDL) level | 12 weeks
  It will be assessed for each pregnant women in the three groups before and after the end of the treatment procedures.The blood samples will be collected after fasting for 9-12 hours. Participants will be asked to lie in half lying position with well supported back and arm, the antecubital area will be cleaned with alcohol. Blood sample of about 5cm will be drawn in the morning (at 8 clock) range between 7and 25 micrograms per deciliter (mcg-dl). Blood sample will be using disposable syringe and collected in sterilized tube.
Assessment of serum high-density lipoprotein (HDL) level | 12 weeks
  It will be assessed for each pregnant women in the three groups before and after the end of the treatment procedures.The blood samples will be collected after fasting for 9-12 hours. Participants will be asked to lie in half lying position with well supported back and arm, the antecubital area will be cleaned with alcohol. Blood sample of about 5cm will be drawn in the morning (at 8 clock) range between 7and 25 micrograms per deciliter (mcg-dl). Blood sample will be using disposable syringe and collected in sterilized tube.

SECONDARY OUTCOMES:
Assessment of level of stress and anxiety | 12 weeks
  Visual analogue scale (VAS) will be used to assess the level of stress and anxiety for each pregnant woman in the three groups. VAS is a straight line; its ends are defined as the extreme limits of stress, with 0 indicates no stress and anxiety, while 10 indicates maximum stress and anxiety. The pregnant woman will select and marks on the line the suitable description of her stress level before and after the end of the treatment course.
Assessment of serum cortisol level | 12 weeks
  It will be assessed for each pregnant women in the three groups before and after the end of the treatment procedures.The blood samples will be collected after fasting for 9-12 hours. Participants will be asked to lie in half lying position with well supported back and arm, the antecubital area will be cleaned with alcohol. Blood sample of about 5cm will be drawn in the morning (at 8 clock) range between 7and 25 micrograms per deciliter (mcg-dl). Blood sample will be using disposable syringe and collected in sterilized tube.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Mohamed Eldeeb, PhD, Study Chair — Professor, Cairo university; Doaa A. Osman, PhD, Study Director — Assistant Professor, Cairo University; Hossam E. Hussein, PhD, Study Director — Professor, Al-Azhar University
Locations (1):
- Cairo University, Giza, Egypt